CLINICAL TRIAL: NCT00890669
Title: Treadmill Walking Training With Additional Body Load Improves Quality of Life in Subjects With Parkinson's Disease
Brief Title: Treadmill Training and Quality of Life in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Nadiesca Taisa Filippin, Universidade Federal de São Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 234/07; CEP/UFSCar
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Parkinson's Disease
Keywords: treadmill training; body load; quality of life; Parkinson's disease; Motor Symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD Group (Experimental): Nine subjects with idiopathic PD, previously diagnosed by one specialist physician participated in this study.
  Interventions: Other: Treadmill walking training with additional body load

INTERVENTIONS:
Other: Treadmill walking training with additional body load — The training program was divided into three phases (A1-B-A2):
  * treadmill training with additional body load (A1),
  * control condition (conventional physical therapy group) (B). and
  * treadmill training with additional body load again (A2).
  Each phase lasted six weeks, totaling 18 weeks. Both evaluations and training were performed during on-phase of the medication cycle.

SUMMARY:
Parkinson's disease (PD) causes motor and non-motor impairments that affect the quality of life of the subjects. The purpose was to assess the effects of treadmill walking training with additional body load on the quality of life and motor symptoms of the subjects with PD.

Methods: Nine subjects with PD, Hoehn and Yahr stages 2 through 3, not demented and with capability to ambulate independently voluntarily participate in this study. The training program was divided into three phases (A1-B-A2): treadmill training with additional body load (A1), control condition (conventional physical therapy group) (B) and treadmill training with load again (A2). Each phase lasted six weeks. The quality of life and motor symptoms were assessed by PDQ-39 and UPDRS, respectively. Both evaluations and training were performed during on-phase of the medication cycle.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr (H-Y) stages 2 through 3
* Absence of dementia (Mini-Mental Status Examination - MMSE, defined according to educational level)
* Capacity to ambulate independently for at least 10 meters

Exclusion Criteria:

* Change medication (dopaminergic) during the study period
* Use treadmill for at least six months prior to the study
* Other neurologic problems or musculoskeletal, cardiovascular and respiratory disease or uncorrected visual deficit that could represent risk and interfere in the accomplishment of the training

Ages: 51 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The quality of life was measured through Parkinson Disease Questionnaire (PDQ-39). | 4 times, once before treatment, and 3 after each treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Nadiesca T Filippin, MSc, Principal Investigator — Universidade Federal de Sao Carlos; Rosana Mattioli, PhD, Study Chair — Universidade Federal de Sao Carlos; Paula H Lobo da Costa, PhD, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil